CLINICAL TRIAL: NCT00432588
Title: Comparing the Effect of Vaginal Misoprostol With Dinoprostone in Term Pregnancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hormozgan University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Misoprostol vs Dinoprostone
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-02

CONDITIONS: Preeclampsia; Fetal Death; Fetal Membranes, Premature Rupture
Keywords: IUFD; POSTTERM; ROM
MeSH Terms: conditions — Pre-Eclampsia; Fetal Death; Fetal Membranes, Premature Rupture | interventions — Misoprostol; Dinoprostone

INTERVENTIONS:
Drug: misoprostol
Drug: dinoprostone

SUMMARY:
Hypothesis (H0): Labor duration and obstetric complications are not significantly different in the three groups (misoprostol-dinoprostone-oxytocin).

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Singleton
* Vertex
* Bishop score below 6

Exclusion Criteria:

* History of drug reaction
* Medical disease
* IUGR
* Oligohydramnios
* Vaginal bleeding
* Fetal anomaly
* Uterine scar

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mitra Ahmad Soltani, Principal Investigator — Hormozgan University of Medical Sciences; Minoo Rajaee Lari, Perinatologist - Obs and Gyn, Study Chair — Department of Obs and Gyn - HUMS
Locations (1):
- Shariaty Maternity Hospital, Tehran, Iran

REFERENCES:
- See also: Related Info — http://www.rcog.org.uk